CLINICAL TRIAL: NCT01428843
Title: A Controlled, Randomised, Double-blind, Multicenter Study, Comparing Ferrisat Versus Placebo in Anemia Associated to Inflammatory Bowel Disease During Anti-TNF Therapy
Brief Title: Comparison of Ferrisat vs Placebo in Anemia Associated to Inflammatory Bowel Disease During Anti-TNF Therapy
Acronym: FER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GETAID 2009-2; 2009-011316-38 (EudraCT Number)
Record Dates: First submitted 2011-08-30; First posted 2011-09-05 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Inflammatory Bowel Disease
Keywords: Inflammatory Bowel Disease; Anemia; Anti-TNF alpha theray; Ferrisat perfusion
MeSH Terms: conditions — Inflammatory Bowel Diseases; Anemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferrisat (Active Comparator): Infusion of Ferrisat (50mg/ml) at inclusion under usual practices
  Interventions: Drug: FERRISAT
- Placebo (Placebo Comparator): Infusion of placebo at inclusion visit
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: FERRISAT — A single infusion of 50 mg/ml of Ferrisat during inclusion visit.
  Other Names: ACTIVE FERRISAT
  Arms: Ferrisat
Drug: PLACEBO — A single infusion of Glucose 5% solution during inclusion visit
  Other Names: GLUCOSE 5%
  Arms: Placebo

SUMMARY:
Anemia is the the most frequently extradigestive symptom for Inflammatory Bowel Disease. This is due to iron deficiency and inflammation.

Most of treatments aim to control inflammation using anti-TNF alpha therapy which should theorically reduce anemia.

The aim of the study is to show that perfusion of iron associated to anti-TNF therapy should reduce anemia and improve quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Crohn's disease or Ulcerative Colitis defined according to the usual endoscopic, histological, and radiological criteria
* Under anti-TNF therapy or indication for starting an anti-TNF therapy
* Anemia defined according to World Health Organization (Hemoglobin under 13g/dl for man and Hemoglobin under 12g/dl for woman)
* Iron deficiency anemia defined as:
* Ferritinemia under 100 if C-Reactive Protein under normal value OR - Ferritinemia between 30 and 100 if C-Reactive Protein above normal value

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Level of hemoglobin | 6 weeks after inclusion
  Efficacy of one-shot perfusion of Ferrisat (Iron supplementation)

SECONDARY OUTCOMES:
Tolerance of Ferrisat | At Inclusion
Improvement of quality of life | 6 weeks after perfusion

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume SAVOYE, PhD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives; Jean-Frédéric COLOMBEL, PhD, Study Director — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives
Locations (18):
- France (18):
  - Chu Amiens, Amiens
  - CHU CAEN, Caen
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - Hopital Bicetre, Le Kremlin-Bicêtre
  - CHRU Lille, Lille
  - Chu Marseille - Hopital Nord, Marseille
  - Chu Nantes, Nantes
  - Hopital Saint Louis, Paris
  - Hopital St Antoine, Paris
  - Hopital Cochin, Paris
  - CHU Bordeaux - Pessac, Pessac
  - CHU LYON, Pierre-Bénite
  - Chu Rennes, Rennes
  - Chu Rouen, Rouen
  - Chu Saint Etienne, Saint-Etienne
  - Chu Toulouse, Toulouse
  - Chu Tours, Tours

REFERENCES:
- [Background] Oldenburg B, Koningsberger JC, Van Berge Henegouwen GP, Van Asbeck BS, Marx JJ. Iron and inflammatory bowel disease. Aliment Pharmacol Ther. 2001 Apr;15(4):429-38. doi: 10.1046/j.1365-2036.2001.00930.x. PMID 11284771
- [Background] Vijverman A, Piront P, Belaiche J, Louis E. Evolution of the prevalence and characteristics of anemia in inflammatory bowel diseases between 1993 and 2003. Acta Gastroenterol Belg. 2006 Jan-Mar;69(1):1-4. PMID 16673554
- [Background] Ormerod TP. Observations on the incidence and cause of anaemia in ulcerative colitis. Gut. 1967 Apr;8(2):107-14. doi: 10.1136/gut.8.2.107. No abstract available. PMID 6022337
- [Result] Wilson A, Reyes E, Ofman J. Prevalence and outcomes of anemia in inflammatory bowel disease: a systematic review of the literature. Am J Med. 2004 Apr 5;116 Suppl 7A:44S-49S. doi: 10.1016/j.amjmed.2003.12.011. PMID 15050885
- [Result] Gasche C, Berstad A, Befrits R, Beglinger C, Dignass A, Erichsen K, Gomollon F, Hjortswang H, Koutroubakis I, Kulnigg S, Oldenburg B, Rampton D, Schroeder O, Stein J, Travis S, Van Assche G. Guidelines on the diagnosis and management of iron deficiency and anemia in inflammatory bowel diseases. Inflamm Bowel Dis. 2007 Dec;13(12):1545-53. doi: 10.1002/ibd.20285. PMID 17985376
- [Result] Gisbert JP, Gomollon F. Common misconceptions in the diagnosis and management of anemia in inflammatory bowel disease. Am J Gastroenterol. 2008 May;103(5):1299-307. doi: 10.1111/j.1572-0241.2008.01846.x. PMID 18477354